CLINICAL TRIAL: NCT00841191
Title: A Phase 1/2, Multiple-Dose, Dose-Escalation Study to Assess the Safety, Efficacy, and Pharmacokinetics of Intravenous CNTO 328, an Anti-Interleukin 6 (IL-6) Monoclonal Antibody, in Subjects With Solid Tumors
Brief Title: A Safety, Efficacy and Pharmacokinetic Study of Siltuximab (CNTO 328) in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015580; CNTO328STM2001; 2008-005180-33
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Ovarian Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms
Keywords: Resistant to anti-EGFR; Interleukin-6; Neoplasms by Histologic Type; Immunologic Factors; Mol Physiological Effects of Drugs; KRAS protein, human; CNTO 328
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms; Colorectal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Neoplasms by Histologic Type | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Siltuximab 2.8 mg/kg (Cohort 1) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody
- Siltuximab 5.5 mg/kg (Cohort 2) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody
- Siltuximab 11 mg/kg (Cohort 3) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody
- Siltuximab 15 mg/kg (Cohort 4) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody
- Siltuximab 15 mg/kg (Expansion Cohort 5) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody
- Siltuximab 15 mg/kg (Ovarian Cancer Cohort 6) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody
- Siltuximab 15 mg/kg (KRAS Mutant Tumors Cohort 7) (Experimental)
  Interventions: Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody

INTERVENTIONS:
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 2.8 milligram per kilogram (mg/kg) will be administered as 1-hour intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) on Day 1, Day 28, Day 42 and Day 56
  Other Names: Siltuximab
  Arms: Siltuximab 2.8 mg/kg (Cohort 1)
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 5.5 mg/kg will be administered as 1-hour intravenous infusion on Day 1, Day 28, Day 42 and Day 56
  Other Names: Siltoximab
  Arms: Siltuximab 5.5 mg/kg (Cohort 2)
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 11 mg/kg will be administered as 1-hour intravenous infusion on Day 1, Day 28, Day 49 and Day 70
  Other Names: Siltuximab
  Arms: Siltuximab 11 mg/kg (Cohort 3)
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 15 mg/kg will be administered as 1-hour intravenous infusion on Day 1, Day 28, Day 49 and Day 70
  Other Names: Siltuximab
  Arms: Siltuximab 15 mg/kg (Cohort 4)
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 15 mg/kg will be administered as 1-hour intravenous infusion once every 21 days for up to a total of 231 days
  Other Names: Siltuximab
  Arms: Siltuximab 15 mg/kg (Expansion Cohort 5)
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 15 mg/kg will be administered as 1-hour intravenous infusion once every 21 days for up to a total of 231 days to participants with ovarian cancer.
  Other Names: Siltuximab
  Arms: Siltuximab 15 mg/kg (Ovarian Cancer Cohort 6)
Drug: CNTO 328; Anti-interleukin-6 monoclonal antibody — Siltuximab 15 mg/kg will be administered as 1-hour intravenous infusion once every 21 days for up to a total of 231 days to participants with tumors harboring Kirsten rat sarcoma viral oncogene homolog (KRAS) mutations or pancreatic cancer, or non-small cell lung cancer (NSCLC), colorectal cancer (CRC), or head and neck (H&N) cancer that were refractory or resistant to anti-epidermal growth factor receptor (EGFR) therapy
  Other Names: Siltuximab
  Arms: Siltuximab 15 mg/kg (KRAS Mutant Tumors Cohort 7)

SUMMARY:
The purpose of this study is to determine the recommended dose of siltuximab monotherapy, in participants with solid malignant (cancerous) tumors (a mass in a specific area) and to estimate the clinical benefit of siltuximab monotherapy in participants with ovarian cancer and with Kirsten rat sarcoma viral oncogene homolog (KRAS) mutant tumors.

DETAILED DESCRIPTION:
This is a 2-part, Phase 1/2, open-label (all people know the identity of the intervention), multiple-dose and dose-escalation study of intravenous (directly into a vein) siltuximab in participants with malignant solid tumors. The study tests the safety and effectiveness of the experimental drug, siltuximab, in participants with advanced cancer (abnormal tissue that grows and spreads in the body). This study also tests how siltuximab is cleared from the body and how the body reacts to it. For this reason blood tests will be performed and some characteristics of the tumor will be analyzed. Siltuximab will be given by intravenous infusion (a fluid or a medicine delivered into a vein by way of a needle) over 1 hour. In Phase 1 (Cohort 1-4) doses will be administered in a range of 2.8-15 milligram per kilogram (mg/kg). Cohort 5 of Phase 1 will receive the recommended dose and schedule as determined from Cohort 1-4. Participants in Phase 1 (Cohort 1-4) will receive 4 administrations of siltuximab over a 10-13 week period, while participants in Cohort 5 and Phase 2 will receive 12 administrations over a 33 week period. Follow-up visits up to 12 weeks after last dose will be scheduled. Participants may then be contacted for up to 1 year after the last dose for follow-up survival and disease status information. Efficacy will primarily be evaluated as per response evaluation criteria in solid tumors (RECIST) criteria. Participants' safety will be monitored at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologic (pertaining to body tissues) or cytologic (pertaining to cells) documentation of malignancy (cancer or other progressively enlarging and spreading tumor) as follows: malignant solid tumors (Cohort 1-4 only); Cohorts 5 and Phase 2: epithelial (tissue covering outer layers of most body organs and parts) ovarian cancers (abnormal tissue growth) that have progressed on or after standard therapy, or for which there is no effective therapy or platinum resistant and taxane resistant, defined as progression on or within 6 months of completing therapy with taxane and platinum either alone or in combination (unless contraindications for taxane or platinum exist), and for which there is no effective therapy, or participants with known KRAS mutant tumors or pancreatic cancer, or non-small cell lung cancer (NSCLC), colorectal cancer (CRC) or head and neck (H&N) cancer that are refractory or resistant to anti-epidermal growth factor receptor (EGFR) therapy and all participants must have received at least 1 line of standard chemotherapy
* Eastern cooperative oncology group (ECOG) performance status score less than or equal to 2
* Participants must have recovered from reversible toxicity (any harmful effect of a drug or poison) of previous treatment to less than or equal to grade 1 or an acceptable baseline
* Women of child bearing potential must have a negative pregnancy test at screening
* Cohort 5 and Phase 2 cohorts must have evaluable or measurable disease (defined by response evaluation criteria in solid tumors [RECIST], as applicable)

Exclusion Criteria:

* Received any prior systemic therapy or had major surgery for the cancer under study within 4 weeks (in the case of nitrosoureas and mitomycin C within 6 weeks) prior to first siltuximab administration
* Prior anti-interleukin 6 (IL-6) targeted therapy
* Serious concurrent illness or history of uncontrolled heart disease such as: unstable angina (chest pain due to decreased oxygen being supplied to the heart), congestive heart failure (failure of the heart resulting in fluid build-up in the lungs, other body tissues, or both), myocardial infarction (heart attack) within preceding 12 months, clinically significant rhythm or conduction abnormality
* Participants with known allergies (over sensitivity to a substance) or clinically significant reactions to murine, chimeric, or human proteins
* Any uncontrolled medical condition, including the presence of laboratory abnormalities, that places the participant at unacceptable risk by participating in the study or confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2009-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Clinical Benefit Response (CBR) | Baseline until disease progression or withdrawal of consent, assessed every 9 weeks up to Week 4 after last dose administration
  The CBR is a confirmed complete response (CR), partial response (PR), or stable disease (SD) lasting at least for 6 weeks as per response evaluation criteria in solid tumors (RECIST) criteria. CR: disappearance of all target and non-target lesions and normalization of tumor marker level; PR: at least 30 percent decrease in sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since treatment started.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Response | Baseline until disease progression or withdrawal of consent, assessed every 9 weeks up to Week 4 after last dose administration
  Overall response is defined as a confirmed CR or PR using RECIST criteria. CR is defined as disappearance of all target lesions and non-target lesions and normalization of tumor marker level, and PR is defined as at least 30 percent decrease in sum of the LD of target lesions, taking as reference the baseline sum LD.
Number of Participants With Tumor Marker Response | Baseline until disease progression or withdrawal of consent, assessed every 9 weeks up to Week 4 after last dose administration
  According to gynecologic cancer intergroup criteria (GCIC), tumor marker response is defined as at least a 50 percent reduction in tumor marker which must be confirmed and maintained for at least 4 weeks. Tumor marker response is assessed using cancer antigen (CA-125), carcinoembryonic antigen (CEA), CA-19.9 and other markers as available
Percentage of Participants With Hemoglobin (Hb) Response | Baseline up to Week 4 after last dose administration
  The Hb response is defined by an increase of at least 1 gram per deciliter (g/dL) over baseline observed at least once in the absence of transfusion or erythropoietin stimulating agents.
Progression Free Survival (PFS) | Baseline until disease progression or death, assessed every 9 weeks up to Week 4 after last dose administration
  The PFS is the time interval between first administration of siltuximab and the first documented sign of progression (at least a 20 percent increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new target or non-target lesions as per RECIST) or death, whichever occurs first.
Overall Survival (OS) | From first dose administration until death, assessed every 3 months up to 12 months after last dose administration
  The OS is the interval between first administration of siltuximab and the participant's death from any cause.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | Baseline up to 4 weeks after last dose administration
  The EORTC QLQ-C30 is used to measure physical function, general health, and global health, as well as participant-reported impression of global quality of life. Symptoms in the scale include: fatigue, pain, and sleep disturbance. It contains 28 items scored using a Likert scale from 1 (not at all) to 4 (very much). 2 additional items are scored from 1 (very poor) to 7 (excellent). Total score ranges from 30-126 with higher score indicating better level of functioning or greater degree of symptoms.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-OV28) Score at Week 4 After Last Dose Administration | Baseline and Week 4 after last dose administration
  The EORTC QLQ-OV28 covers side effects of therapy; activity limitation attributable to disease; hormonal symptoms; body image; difficulty with specific bodily functions; and sexual functioning. It contains 28 items scored using a Likert scale from 1 (not at all) to 4 (very much) with a recall period of the past week or, in the final segment, the past 4 weeks. Total score ranges from 28-112 with higher score indicating better level of functioning or greater degree of symptoms.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  Area under the serum concentration versus time curve from time zero to infinity with extrapolation of the terminal phase will be calculated; samples for the determination of siltuximab serum concentration will be collected from 0 hour (h) (pre-dose) to 24h (post-dose) on Day (D) 1 up to Week 12 (Wk12) after last dose administration for all cohorts.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUC[0-t]) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  Area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (AUC[0-t]) was calculated.
Minimum Observed Serum Concentration at Steady-State (Cmin,ss) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  The Cmin,ss is the minimum observed serum concentration during a dosing interval at steady-state (time at which serum concentration does not change with time).
Maximum Observed Serum Concentration (Cmax) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  The Cmax is the maximum observed serum concentration of siltuximab.
Terminal Elimination Half Life (t1/2) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  Terminal elimination half-life is the time measured for the serum concentration to decrease to half value.
Total Systemic Clearance (CL) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  Total systemic CL is calculated by dividing the dose by area under the curve from time 0 to extrapolated infinite time (AUCinf).
Volume of Distribution at Steady State (Vss) | Cohort1-4:0,1,4,6,24h post-dose on D1,8,15,22; D1 of extended treatment; Cohort1,2:0,1h post-dose on D28,42,56; Cohort3,4:D28,49,70; Cohort5-7:0,1,2h post-dose on D1,8,15; 0,1h post-dose on D21,42,63,84,105,168,231; up to Wk12 after last dose (Cohort1-7)
  The Vss is calculated by multiplying mean residence time (MRT) with systemic clearance (CL). MRT is the time when 63.2 percent of an intravenous dose has been eliminated after single dose administration.
Percent Change From Baseline in C-Reactive Protein (CRP) Level | Baseline; Day (D) 1,8,15 (post-dose) for cohort 1 to 7; Day 22 (post-dose), 28 (pre-dose) for cohort 1 to 4; Day 42,56 (pre-dose) for cohort 1, 2; Day 49,70 (pre-dose) for cohort 3, 4; Day 21,42,63,84,105,126,147,168,189,210 (pre-dose) for cohort 5 to 7
  The CRP levels are determined using high sensitive CRP assay and percent change from baseline is calculated at each time point.
Percent Change From Baseline in Inflammatory Cytokines Level | Baseline; Day 8 and 15 (post-dose) for cohort (C) 1 to 7; Day 22 (post-dose) and 28 (pre-dose) for cohort 1 to 4; Day 42 and 56 (pre-dose) for cohort 1 and 2; Day 49 and 70 (pre-dose) for cohort 3 and 4; Day 21, 42 and 63 (pre-dose) for cohort 5 to 7
  Percent change from baseline in the levels of inflammatory (pertaining to pain, redness and swelling) markers for interferon gamma (IFN-g), interleukin 1 beta (IL1b), IL-2, IL-5, IL-8, IL10, IL12, and tumor necrosis factor alpha (TNFa) is calculated.
Percent Change From Baseline in the Angiogenesis Related Factors Level | Baseline; Day 8 and 15 (post-dose) for cohort 1 to 7; Day 22 (post-dose) and 28 (pre-dose) for cohort 1 to 4; Day 42 and 56 (pre-dose) for cohort 1 and 2; Day 49 and 70 (pre-dose) for cohort 3 and 4; Day 21, 42 and 63 (pre-dose) for cohort 5 to 7
  Percent change from baseline in the level of markers associated with angiogenesis related factors (vascular endothelial growth factor [VEGF], vascular endothelial growth factor receptor [VEGFR], and basic fibroblast growth factor [bFGF]) is calculated.
Percent Change From Baseline in Interleukin 6 Receptor (IL-6R) Subunits Level | Baseline; Day 8 and 15 (post-dose) for cohort 1 to 7; Day 28 (pre-dose) for cohort 1 to 4; Day 42 and 56 (pre-dose) for cohort 1 and 2; Day 49 and 70 (pre-dose) for cohort 3 and 4; Day 21, 42 and 63 (pre-dose) for cohort 5 to 7
  Percent change from baseline in the level of ligand-binding subunit of the IL-6R, soluble GP80 (sGP80) and signal-transducing subunit of the IL-6R, soluble GP130 (sGP130) is calculated.
Number of Participants Assessed Positive for Antibodies to Siltuximab | Day 1 (pre-dose) up to Week 12 after last dose administration
  Number of participants who are tested positive for antibodies (type of protein that helps to protect the body against foreign matter, such as bacteria and viruses) to siltuximab is reported.
Percent Change From Baseline in Hepcidin Level | Baseline; Day 8 and 15 (post-dose) for cohort 1 to 7; Day 22 (post-dose) and 28 (pre-dose) for cohort 1 to 4; Day 42 and 56 (pre-dose) for cohort 1 and 2; Day 49 and 70 (pre-dose) for cohort 3 and 4; Day 21, 42 and 63 (pre-dose) for cohort 5 to 7
  Hepcidin is a liver-produced iron-regulatory peptide hormone (substance made by a gland in the body that regulates another part of the body) that is implicated in anemia (decreased number of red blood cells) of inflammation (pain, redness and swelling). Percent change from baseline in hepcidin (marker of anemia and iron metabolism) level is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (12):
- United States (2):
  - Philadelphia, Pennsylvania
  - Houston, Texas
- Belgium (2):
  - Brussels
  - Wilrijk
- France (3):
  - Caen
  - Lyon
  - Villejuif
- Spain (2):
  - Barcelona
  - Madrid
- United Kingdom (3):
  - Birmingham
  - Edinburgh
  - Southampton

REFERENCES:
- See also: A Phase 1/2, Multiple-dose, Dose-escalation Study to Assess the Safety, Efficacy, and Pharmacokinetics of Intravenous CNTO 328, an Anti-Interleukin 6 (IL-6) Monoclonal Antibody, in Subjects with Solid Tumors — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=191&filename=CR015580_CSR.pdf